CLINICAL TRIAL: NCT00861796
Title: A Multi-center, Inpatient and Ambulatory, Phase 2, Double Blind, Randomized, Placebo-controlled Proof of Concept Study of CYR-101 in Patients With DSM-IV Schizophrenia
Brief Title: Study of CYR-101 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyrenaic Pharmaceuticals (Industry)
Responsible Party: Lorenzo Pellegrini, Cyrenaic Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYR-101C01
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CYR-101
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CYR-101 — Experimental arm
  Arms: 1
Drug: Placebo — Placebo comparator
  Arms: 2

SUMMARY:
This Phase II study will test whether CYR-101, a CNS-active compound with novel pharmacological profile and devoid of dopamine D2 receptor binding properties, is efficacious when administered orally in the management of patients with a diagnosis of DSM-IV schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 65 years of age, inclusive
* Female patients must test negative for pregnancy and, if of childbearing potential, must be using a medically accepted means of contraception.
* Patients must have a diagnosis of Schizophrenia or schizo-affective disorders as defined in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revised (DSM-IV TR, APA 2000) (Disorganised, 295.10; Catatonic, 295.20; Paranoid, 295.30; Residual, 295.60; or Undifferentiated, 295.90) and confirmed by the Structured Clinical Interview for DSM-IV (SCID).
* Patients must meet the following psychopathologic severity criteria at screening: Positive and Negative Syndrome Scale (PANSS) total score, of at least 60.
* Patients must receive a rating of 4 (moderately ill) or greater on the Clinical Global Impression-Severity (CGI-S) scale at screening.
* Patients in whom, in the opinion of the investigator, a switch to another antipsychotic medication or initiation of an antipsychotic medication is indicated.
* Patients must be considered reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol.
* Patients must be able to understand the nature of the study and have given their own informed consent.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Have received treatment with a drug that has not received regulatory approval for any indication within 30 days prior to screening.
* Patients in whom treatment with CYR-101, or placebo, as specified in this protocol, is relatively or absolutely clinically contraindicated.
* Patients who have a history of an inadequate response, in the opinion of the investigator, to 2 or more adequate antipsychotic medication trials of at least 8 weeks duration in the past 12 months prior to screening.
* Patients who require concomitant treatment with any other medication with primary central nervous system activity, other than certain allowed medications as specified in Study Protocol.
* Patients receiving treatment with depot antipsychotic medication within 1 dosing interval, minimum of 4 weeks, prior to screening.
* Actively suicidal (for example any suicide attempts within the past month or any current suicidal intent including plan) in the opinion of the investigator or a score of 4 or greater on Item 10 of the Montgomery-Asberg Depression Rating Scale (MADRS).
* DSM-IV diagnosis of substance dependence or substance abuse (except nicotine and caffeine) within the 6 months prior to screening.
* Diagnosis of substance-induced psychosis by DSM-IV criteria within 7 days of screening (or at any time during the study).
* Patients with current heteroaggressive behavior.
* Female patients who are pregnant, nursing, or who intend to become pregnant within 30 days of completing the study.
* Have increased risk of seizures as evidenced by a history of: one or more seizures (except childhood febrile seizure), history of electroencephalogram (EEG) with epileptiform activity, history of stroke; surgery to the cerebral cortex; or head trauma with loss of consciousness. NOTE: patients with a history of childhood febrile seizure may be enrolled in this study.
* Patients who have had electroconvulsive therapy (ECT) within 3 months of screening visit or who will have ECT at any time during the study.
* Test HIV positive.
* Test positive for Hepatitis C antibody or Hepatitis B surface antigen (HBsAg). Patients with positive Hepatitis B core antibody test and negative HBsAg may be included in the study if aminotransferase levels (ALT/SGPT and AST/SGOT) do not exceed 1.5 times upper limit of normal (ULN).
* Alanine transaminase/serum glutamic-pyruvic transaminase (ALT/SGPT) values >1.5 times ULN of the performing laboratory, or total bilirubin values >2 times the ULN or concomitant ALT/SGPT values >1.5 times the ULN and total bilirubin values >1.5 times the ULN at screening.
* Patients with acute, serious, or unstable medical conditions, including (but not limited to) inadequately controlled diabetes (hemoglobin A1c (HbA1c) >8%), severe hypertriglyceridemia (fasting triglycerides >5.6 mmol/L, recent cerebrovascular accidents, serious acute systemic infection or immunologic disease, unstable cardiovascular disorders (including ischemic heart disease), malnutrition, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, or haematologic diseases.
* Prolactin level at screening visit of greater than 200 ng/mL (or 200mg/L).
* A diagnosis of Parkinson's disease, dementia-related psychosis, or related disorders. If a patient has a past misdiagnosis of Parkinson's disease, dementia-related psychosis, or related disorders, the investigator will need to contact the Clinical Research Physician prior to enrolment.
* Patient with current clinically significant cardiovascular disease.
* History of syncopal events due to cardiovascular abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Global PANSS score and sub-scores | one month (28 days +/- 2 days)

SECONDARY OUTCOMES:
PANSS total score and sub-scores | Three months (84 days +/- 2 days)
CGI-S, DAI-10, PSQI, BACS, MADRS, HAMA. | three months (84 days +/- 2 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nancy (CHU), Toul, France